CLINICAL TRIAL: NCT01076972
Title: Drug Use Investigation of Kaletra
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: PMOS-JAP-00-001
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-01

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lopinavir/ritonavir group: All patients in this non-interventional, post-marketing observational study, who were prescribed lopinavir/ritonavir (Kaletra) in accordance with the local Prescribing Information for the treatment of HIV infection.
  Interventions: Drug: Lopinavir/ritonavir (Kaletra)

INTERVENTIONS:
Drug: Lopinavir/ritonavir (Kaletra) — Lopinavir/ritonavir evaluated separately in patients who were naive to previous antiretroviral treatment and those who were not.
  Other Names: Lopinavir/ritonavir; Kaletra

SUMMARY:
This non-interventional, post-marketing observational study was conducted to obtain data, such as safety and effectiveness, from the use of lopinavir/ritonavir (Kaletra) in clinical practice and investigate the necessity to conduct a follow-up post-marketing clinical study in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All patients prescribed Kaletra for the treatment of HIV are eligible for this survey.

Exclusion Criteria:

* Contraindications according to the Package Insert:

  * Patients with a history of hypersensitivity to any ingredient of Kaletra
  * Patients who are receiving pimozide, cisapride, ergotamine tartrate, dihydroergotamine mesylate, ergometrine maleate, methylergometrine maleate, midazolam, triazolam, vardenafil hydrochloride hydrate, boriconazol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1184 (Actual)
Dates: Start 2000-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yo Hoshino, Study Director — Abbott Japan Co.,Ltd
Locations (29):
- Japan (29):
  - Site Reference ID/Investigator# 36516, Aichi
  - Site Reference ID/Investigator# 36517, Aichi
  - Site Reference ID/Investigator# 36518, Chiba
  - Site Reference ID/Investigator# 36519, Fukuoka
  - Site Reference ID/Investigator# 36521, Fukuoka
  - Site Reference ID/Investigator# 36522, Hiroshima
  - Site Reference ID/Investigator# 36523, Hokkaido
  - Site Reference ID/Investigator# 36524, Hyōgo
  - Site Reference ID/Investigator# 36525, Kanagawa
  - Site Reference ID/Investigator# 36526, Kyoto
  - Site Reference ID/Investigator# 36622, Miyagi
  - Site Reference ID/Investigator# 36623, Miyagi
  - Site Reference ID/Investigator# 36624, Niigata
  - Site Reference ID/Investigator# 36625, Okayama
  - Site Reference ID/Investigator# 36626, Osaka
  - Site Reference ID/Investigator# 36627, Osaka
  - Site Reference ID/Investigator# 36628, Shizuoka
  - Site Reference ID/Investigator# 36629, Tokyo
  - Site Reference ID/Investigator# 36630, Tokyo
  - Site Reference ID/Investigator# 36631, Tokyo
  - Site Reference ID/Investigator# 36632, Tokyo
  - Site Reference ID/Investigator# 36633, Tokyo
  - Site Reference ID/Investigator# 36634, Tokyo
  - Site Reference ID/Investigator# 36635, Tokyo
  - Site Reference ID/Investigator# 36636, Tokyo
  - Site Reference ID/Investigator# 36637, Tokyo
  - Site Reference ID/Investigator# 36638, Tokyo
  - Site Reference ID/Investigator# 36639, Tokyo
  - Site Reference ID/Investigator# 5342, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir Group
Started | 1184
Completed | 1184
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 1184
Age Continuous [Mean (Standard Deviation); unit: years] | 39.7 (11.0)
Age, Customized [Number; unit: participants]
  <=14 years | 4
  Between 15 and 64 years | 1155
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 1078
Region of Enrollment [Number; unit: participants]
  Japan | 1184

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Patients With Adverse Drug Reactions
Description: Number of patients with adverse drug reactions, defined as adverse events for which the causal relationship with Kaletra was something other than "not related" by the investigator (i.e., "probable," "possible," or "unclear"), that occurred in ≥ 5% of patients. Adverse drug reactions are reported by preferred term and inclusive of all those reported at each visit. Although a patient may experience a particular preferred term more than once, each patient was counted only once for each preferred term.
Time Frame: During the course of the survey period up to Year 8
Population: Available data for all patients were included.
Measure: Number; unit: participants
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 1184
participants
  Any adverse drug reaction | 649
  Hypertriglyceridaemia | 67
  Hyperlipidaemia | 211
  Diarrhoea | 130
  Nausea | 72
  Blood triglycerides increased | 99

2. Primary Outcome: Cluster of Differentiation 4 Lymphocyte Count (CD4)
Description: The evolution of patients' CD4-positive (CD4+) T-lymphocyte counts after starting treatment with Kaletra was assessed by measuring the number of CD4+ cells at baseline and each subsequent study visit. CD4+ counts are reported as the number of CD4+ cells per cubic millimeter (cmm) and presented by the mean at each visit. Only observed cases were included in analyses; no data were imputed. n = xx, xx is the number of patients naive to previous antiretroviral treatment and those that were not who had CD4+ T-cell counts available for analysis at each study visit.
Time Frame: Baseline (Month 0), every 3 months thereafter up to Month 12 and every year thereafter up to Year 8 (Month 96) during the course of the survey period
Population: Available data at each visit for each subgroup of patients who had not received and received prior antiretroviral drug therapy were included in the analyses. Data for patients for whom either baseline or treatment data were missing for a given visit were excluded from the analysis for that visit.
Measure: Mean (Standard Deviation); unit: cells per cubic millimeter
Groups:
- Lopinavir/Ritonavir: Treatment-Naive: The subgroup of patients who had not received prior antiretroviral drug therapy. Data for patients for whom either baseline data or data during treatment were missing for a given time point were excluded from the analysis for that time point. Of the 1184 total enrolled patients, 416 patients had baseline data and efficacy data for this outcome measure, and were therefore included in the analysis.
- Lopinavir/Ritonavir: Treatment-Experienced: The subgroup of patients who have received prior antiretroviral drug therapy. Data for patients for whom either baseline data or data during treatment were missing for a given time point were excluded from the analysis for that time point. Of the 1184 total enrolled patients, 420 patients had baseline data and efficacy data for this outcome measure, and were therefore included in the analysis.
Arm/Group | Lopinavir/Ritonavir: Treatment-Naive | Lopinavir/Ritonavir: Treatment-Experienced
Number analyzed (Participants) | 416 | 420
cells per cubic millimeter
  Baseline (Month 0 [n = 416, 420]) | 125.0 (123.5) | 290.6 (224.6)
  Month 3 (n = 315, 283) | 257.2 (170.8) | 342.9 (230.5)
  Month 6 (n = 288, 252) | 275.9 (175.4) | 366.4 (227.0)
  Month 9 (n = 223, 238) | 311.1 (175.1) | 385.0 (224.3)
  Month 12 (Year 1 [n = 201, 233]) | 329.9 (178.6) | 410.4 (214.7)
  Year 2 (n = 146, 190) | 419.4 (201.1) | 437.4 (224.2)
  Year 3 (n = 106, 150) | 455.6 (202.4) | 481.5 (255.4)
  Year 4 (n = 69, 99) | 475.2 (209.6) | 526.6 (296.4)
  Year 5 (n = 40, 73) | 535.1 (248.0) | 496.2 (228.7)
  Year 6 (n = 25, 42) | 577.1 (241.9) | 569.7 (287.0)
  Year 7 (n = 3, 17) | 602.0 (156.1) | 597.7 (224.2)
  Year 8 (n = 0, 3) | NA (NA) — No data were recorded for any patients at this visit. | 493.7 (414.8)

3. Primary Outcome: Mean Number of Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) Copies Per Milliliter (mL) Using a Logarithmic (Base 10) Transformation at Each Visit
Description: Number of HIV RNA copies per mL is presented by the mean per visit for patients that were naive to previous antiretroviral treatment and those that were not. HIV-RNA data reported as < 400 copies/mL were considered 399 copies/mL in calculations. The mean and standard deviation of HIV-RNA levels were thus calculated after logarithmic (base 10) transformation (log10 399 is 2.6). Only observed cases were included in analyses; no data were imputed. n = xx, xx is the number of treatment-naive, treatment-experienced participants who had CD4+ T-cell counts available for analysis at each study visit.
Time Frame: as for outcome 2
Population: Available data at each visit for each subgroup of patients who had not received and who had received prior antiretroviral drug therapy were included in the analyses. Data for patients for whom either baseline data or treatment data were missing for a given visit were excluded from the analysis for that visit.
Measure: Mean (Standard Deviation); unit: copies/mL
Groups:
- Lopinavir/Ritonavir: Treatment-experienced: The subgroup of patients who have received prior antiretroviral drug therapy. Data for patients for whom either baseline data or data during treatment were missing for a given time point were excluded from the analysis for that time point. Of the 1184 total enrolled patients, 418 patients had baseline data and efficacy data for this outcome measure, and were therefore included in the analysis.
Arm/Group | Lopinavir/Ritonavir: Treatment-Naive | Lopinavir/Ritonavir: Treatment-experienced
Number analyzed (Participants) | 416 | 418
copies/mL
  Baseline (Month 0 [n = 416, 418]) | 4.9 (0.8) | 3.5 (1.1)
  Month 3 (n = 315, 280) | 2.7 (0.4) | 2.8 (0.5)
  Month 6 (n = 288, 253) | 2.7 (0.3) | 2.8 (0.6)
  Month 9 (n = 224, 238) | 2.6 (0.3) | 2.8 (0.5)
  Month 12 (Year 1 [n = 203, 230]) | 2.7 (0.4) | 2.8 (0.6)
  Year 2 (n = 145, 190) | 2.7 (0.3) | 2.7 (0.5)
  Year 3 (n = 107, 147) | 2.6 (0.1) | 2.7 (0.4)
  Year 4 (n = 70, 99) | 2.6 (0.1) | 2.7 (0.4)
  Year 5 (n = 39, 72) | 2.7 (0.3) | 2.8 (0.5)
  Year 6 (n = 25, 41) | 2.7 (0.3) | 2.6 (0.3)
  Year 7 (n = 3, 17) | 2.6 (0.0) | 2.8 (0.6)
  Year 8 (n = 0, 3) | NA (NA) — No data were recorded for any patients at this visit. | 2.6 (0.0)

4. Primary Outcome: Number of Patients Included in Each Center for Disease Control and Prevention (CDC) Classification Category for HIV-infected Adults and Adolescents
Description: Number of patients in each CDC category at Baseline (last assessment within 30 days prior to first dose of Kaletra) and after treatment. CDC categories defined as: Category A (asymptomatic acute HIV infection), Category B (symptomatic HIV infection; not Categories A and C), Category C (acquired immunodeficiency syndrome [AIDS] indicator status), Class P-0 (children not confirmed for HIV infection), Class P-1 (children with asymptomatic HIV infection), or Class P-2 (children with symptomatic HIV infection).
Time Frame: Baseline (Month 0) and following last treatment dose during the course of the survey period
Population: Available data for all patients were included.
Measure: Number; unit: participants
Groups:
- Lopinavir/Ritonavir: Baseline Category A: The subgroup of patients who were classified as CDC Category A at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category B: The subgroup of participants who were classified as CDC Category B at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category C: The subgroup of patients who were classified as CDC Category C at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category P-0: The subgroup of participants who were classified as CDC Category P-0 at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category P-1: The subgroup of participants who were classified as CDC Category P-1 at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category P-2: The subgroup of participants who were classified as CDC Category P-2 at Baseline (prior to treatment with lopinavir/ritonavir).
- Lopinavir/Ritonavir: Baseline Category Unknown: The subgroup of participants whose CDC classification at Baseline (prior to treatment with lopinavir/ritonavir) was unknown.
Arm/Group | Lopinavir/Ritonavir: Baseline Category A | Lopinavir/Ritonavir: Baseline Category B | Lopinavir/Ritonavir: Baseline Category C | Lopinavir/Ritonavir: Baseline Category P-0 | Lopinavir/Ritonavir: Baseline Category P-1 | Lopinavir/Ritonavir: Baseline Category P-2 | Lopinavir/Ritonavir: Baseline Category Unknown
Number analyzed (Participants) | 378 | 71 | 323 | 0 | 0 | 1 | 411
participants
  Category A after lopinavir/ritonavir treatment | 206 | 0 | 0 |  |  | 0 | 103
  Category B after lopinavir/ritonavir treatment | 2 | 32 | 0 |  |  | 0 | 22
  Category C after lopinavir/ritonavir treatment | 6 | 2 | 191 |  |  | 0 | 86
  Category P-0 after lopinavir/ritonavir treatment | 0 | 0 | 0 |  |  | 0 | 0
  Category P-1 after lopinavir/ritonavir treatment | 0 | 0 | 0 |  |  | 0 | 1
  Category P-2 after lopinavir/ritonavir treatment | 0 | 0 | 0 |  |  | 0 | 0
  Category unknown after treatment | 164 | 37 | 132 |  |  | 1 | 199

ADVERSE EVENTS:
Time Frame: During the course of the survey period up to Year 8.
Description: Adverse drug reactions (ADRs) for Primary Outcome Measure 1, defined as AEs (a) for which the causal relationship with Kaletra was other than 'not related' (including 'unclear') and (b) which occurred in > 5% of patients, were summarized from the list of AEs below. ADRs are inclusive of all such events reported at each visit.
Arm/Group | Lopinavir/Ritonavir Group
Serious Adverse Events (participants affected / at risk) | 189/1184
Other Adverse Events (participants affected / at risk) | 539/1184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir Group (N=1184)
Acute tonsillitis (Infections and infestations) | 1
Amoebic dysentery (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 2
Cryptosporidiosis infection (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis salmonella (Infections and infestations) | 1
Genital herpes (Infections and infestations) | 1
Giardiasis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 10
Influenza (Infections and infestations) | 1
Measles (Infections and infestations) | 1
Meningitis cryptococcal (Infections and infestations) | 2
Meningitis herpes (Infections and infestations) | 1
Neurosyphilis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Pneumonia pneumococcal (Infections and infestations) | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1
Prostatic abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Cytomegalovirus chorioretinitis (Infections and infestations) | 4
AIDS encephalopathy (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 2
Cerebral toxoplasmosis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Mycobacterium avium complex infection (Infections and infestations) | 1
Anogenital warts (Infections and infestations) | 2
Tuberculosis gastrointestinal (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 2
Hepatic amoebiasis (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 5
Extrapulmonary tuberculosis (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 13
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1
Behcet's syndrome (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Immune reconstitution syndrome (Immune system disorders) | 8
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyperlactacidaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Lactic acidosis (Metabolism and nutrition disorders) | 3
Malnutrition (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Eating disorder (Psychiatric disorders) | 1
Emotional disorder (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 2
Mania (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 4
Cerebral infarction (Nervous system disorders) | 4
Convulsion (Nervous system disorders) | 5
Encephalitis (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 3
Guillain-Barre syndrome (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 1
Myelitis (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Paralysis (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Ulcerative keratitis (Eye disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Myocarditis (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Sinus arrest (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Kawasaki's disease (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Intra-abdominal haematoma (Vascular disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 3
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Pancreatitis acute (Gastrointestinal disorders) | 3
Pancreatitis relapsing (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Subileus (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 3
Hepatitis acute (Hepatobiliary disorders) | 1
Hepatitis fulminant (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Osteomalacia (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Calculus urinary (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 3
Epididymitis (Reproductive system and breast disorders) | 1
Fanconi syndrome (Congenital, familial and genetic disorders) | 1
Death (General disorders) | 2
Necrosis (General disorders) | 1
Pyrexia (General disorders) | 1
C-reactive protein increased (Investigations) | 1
Chest X-ray abnormal (Investigations) | 1
Platelet count decreased (Investigations) | 6
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 4
Protein urine present (Investigations) | 1
Transaminases increased (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lopinavir/Ritonavir Group (N=1184)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 77
Hyperlipidaemia (Metabolism and nutrition disorders) | 230
Diarrhoea (Gastrointestinal disorders) | 148
Nausea (Gastrointestinal disorders) | 87
Blood triglycerides increased (Investigations) | 104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.